CLINICAL TRIAL: NCT04795648
Title: Spatial Repellent Products for Control of Vector Borne Diseases
Brief Title: Spatial Repellents for Vector Control
Acronym: AEGIS Mali
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Notre Dame (Other)
Collaborators: S.C. Johnson & Son, Inc. (Industry); fhiClinical (Unknown); Malaria Research and Training Center, Bamako, Mali (Other); Catholic Relief Services (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 20-10-6245
Record Dates: First submitted 2021-03-09; First posted 2021-03-12 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-04

CONDITIONS: Malaria
Keywords: Malaria; Spatial Repellent; Transfluthrin; Vector-borne diseases; Mosquito vectors; Incidence
MeSH Terms: conditions — Malaria; Vector Borne Diseases

STUDY DESIGN:
Intervention Model Description: The study design will be a prospective cluster Randomized Control Trial (cRCT)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Spatial Repellent (Experimental): Transfluthrin
  Interventions: Device: Transfluthrin
- Placebo (Placebo Comparator): Inert ingredients
  Interventions: Device: Placebo

INTERVENTIONS:
Device: Transfluthrin — Passive emanator with formulated transfluthrin
  Arms: Spatial Repellent
Device: Placebo — Passive emanator with formulated inert ingredients
  Arms: Placebo

SUMMARY:
The primary objective of the study is to demonstrate and quantify the protective efficacy of a single Spatial Repellent (SR) product, in reducing malaria infection in a human cohort. The study design will be a prospective cluster Randomized Control Trial (cRCT).

DETAILED DESCRIPTION:
Children ≥ 6 months to < 10 years of age will be enrolled in a single cohort across 60 clusters (30 clusters per treatment arm). The cohort will be followed for 6 months for baseline covariate measurements and 24 months with intervention. Blood samples will be taken once every 4 weeks from all cohort subjects to test for malaria infection and whenever a subject reports a recent history of fever (within previous 48 hours). During follow up of enrolled subjects, study clinicians will have the option to conduct a Hb test for enrolled subjects when they may present signs of anemia to see if they might need additional treatment beyond malaria ACTs (if malaria infection is indicated). Rapid Diagnostic Tests (RDTs) will be used for point-of-care diagnosis of malaria infection with microscopy used to confirm infection status. All positive malaria infections as indicated by either RDT or microscopy, clinical and asymptomatic, will be treated. If a subject has a RDT negative outcome but a positive microscopy diagnosis, follow up treatment for the malaria infection will be provided to the subject within 72hrs of the microscopy read. Cohort subjects who test positive for malaria by either RDT or microscopy, symptomatic or asymptomatic, during both scheduled and unscheduled visits will be treated with ACTs. The incidence of malaria infection will be measured by microscopy and estimated and compared between treatment arms to determine the benefit of using an SR in an area with high, seasonal transmission of malaria.

Entomological endpoints of exposure risk to mosquitoes will also be measured to identify entomological correlates of SR efficacy that may be useful for the evaluation of new SR products. Twenty clusters (10 SR, 10 placebo) will be randomly selected to estimate the impact of the SR on entomological measures of malaria transmission. Within each cluster, light trap collections will be conducted monthly in 10 randomly selected households to assess the impact of SRs on the density of Anopheles mosquitoes indoors. Human landing catches will be done indoors and outdoors in 6 intervention and 6 control clusters (the 12 clusters will remain fixed throughout the study) in four houses (randomly selected) in each cluster for the period of 2 nights (total of 48 houses across both arms) once every quarter (3 months) to determine the effect of SR on the host seeking behavior of mosquitoes.

The SR will be a new formulation of transfluthrin. This active ingredient (AI) is widely used in mosquito coils and other household pest control products. The new formulation is a passive emanator that will release the AI over a period of up to four weeks. The emanator will consist of a pre-treated piece of cellulose acetate, which will be positioned within consenting households according to manufacturer specifications. The SRs and placebos for this study will be designed and manufactured by S.C. Johnson, Inc. USA.

ELIGIBILITY:
Inclusion Criteria:

* Children ≥ 6 months to < 10 years of age
* Children with Hb > 7 g/dL and no signs of known chronic disease or other other serious illness
* Sleeps in cluster ≥ 90% of nights during any given month
* Not participating in another clinical trial investigating a vaccine, drug, medical device, or a medical procedure during the trial
* Provision of informed consent (and/or assent) form (ICF) signed by the parent(s) or guardian

Exclusion Criteria:

* Children < 6 months or ≥ 10 years
* Childrend with Hb <= 7 g/dL with signs of known chronic disease or other serious illness, or Hb <6 g/dL with signs of clinical decompensation
* Sleeps in cluster <90% of nights during any given month
* Participating or planned participation in another clinical trial investigating a vaccine, drug, medical device, or a medical procedure during the trial
* No provision of ICF (and/or assent) signed by the parent(s) or guardian

Ages: 6 Months to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1911 (Actual)
Dates: Start 2021-07-08 (Actual); Primary Completion 2024-03-02 (Actual); Study Completion 2024-03-02 (Actual)

PRIMARY OUTCOMES:
Number of first-time malaria infections during intervention period. | 24 months
  Measured by microscopy in children aged between 6 months to 10 years.

SECONDARY OUTCOMES:
Number of overall new malaria infections during intervention period. | 24 months
  Measured by microscopy in children aged between 6 months to 10 years.
Parasite-species-specific first-time malaria infections. | 24 months
  Measured by microscopy in children aged between 6 months to 10 years.
Parasite-species-specific overall malaria infections. | 24 months
  Measured by microscopy in children aged between 6 months to 10 years.
Number of first-time malaria infections by two age groups (≤ 59 months old; 5 years old to 10 years old). | 24 months
  Measured by microscopy in children aged between 6 months to 10 years.
Number of overall malaria infections by two age groups (≤ 59 months old; 5 years to 10 years old). | 24 months
  Measured by microscopy in children aged between 6 months to 10 years.
Anopheline-human contact (indoor and outdoor) using human biting rate (HBR) as an indicator for all anophelines and by anopheline species. | 24 months
  Measured by human-landing catch (HLC) during 12-h intervals on a quarterly basis during intervention period.
Anopheline parity rate as an indicator of population age structure for all anophelines and by anopheline species. | 24 months
  Measured by mosquito ovarian dissections from a sub-sample of anophelines collected during HLC procedures during intervention period.
Anopheline infectivity using sporozoite rate as an indicator for all anophelines and by anopheline species. | 24 months
  Measured by laboratory detection of sporozoites in mosquito head-preps from a sub-sample of anophelines collected during HLC and/or CDC-light trap procedures during intervention period.
Anopheline infectivity using entomological inoculation rate (EIR) as an indicator for all anophelines and by anopheline species. | 24 months
  Measured by calculating the number of sporozoite-infected anopheline mosquitoes captured per person during intervention period from HLC and/or CDC-light trap procedures.
CDC-light trap indoor density for all anophelines and by anopheline species. | 24 months
  Measured by CDC-light trap collections during 12-h intervals on a monthly basis during intervention period.
Insecticide resistance. | 30 months
  Measured by WHO filter paper test and CDC bottle assays during baseline and intervention period.
Adverse Events and Serious Adverse Events. | 30 months
  Measured by solicited and unsolicited reports during baseline and intervention period. Mean, minimum and maximum frequency and percentage of Adverse Events(AEs) and Severe Adverse Events (SAEs) across clusters among enrolled subjects will be summarized by treatment arm.

CONTACTS AND LOCATIONS:
Overall Officials: John P Grieco, Ph.D., Study Director — University of Notre Dame; Suzanne Van Hulle, M.H.S, Principal Investigator — Catholic Relief Services
Locations (2):
- Mali (2):
  - Catholic Relief Services, Bamako
  - Malaria Research and Training Center (MRTC), University of Bamako, Mali, Bamako

IPD SHARING:
Plan to Share IPD: Yes
Analytical datasets will be anonymized and GPS tag-blurred to remove sensitive information prior to sharing.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: The data and supporting information will be made available 12 months following completion of data analysis and will remain open access in the public domain.
Access Criteria: Open-access repository distributed under the terms of the Creative Commons Attribution (CC-BY) License, which permits unrestricted use, distribution, and reproduction in any medium, provided the original author and source are credited.

REFERENCES:
- [Background] Achee NL, Bangs MJ, Farlow R, Killeen GF, Lindsay S, Logan JG, Moore SJ, Rowland M, Sweeney K, Torr SJ, Zwiebel LJ, Grieco JP. Spatial repellents: from discovery and development to evidence-based validation. Malar J. 2012 May 14;11:164. doi: 10.1186/1475-2875-11-164. PMID 22583679
- [Background] Cisse MB, Keita C, Dicko A, Dengela D, Coleman J, Lucas B, Mihigo J, Sadou A, Belemvire A, George K, Fornadel C, Beach R. Characterizing the insecticide resistance of Anopheles gambiae in Mali. Malar J. 2015 Aug 22;14:327. doi: 10.1186/s12936-015-0847-4. PMID 26296644
- [Background] Fanello C, Petrarca V, della Torre A, Santolamazza F, Dolo G, Coulibaly M, Alloueche A, Curtis CF, Toure YT, Coluzzi M. The pyrethroid knock-down resistance gene in the Anopheles gambiae complex in Mali and further indication of incipient speciation within An. gambiae s.s. Insect Mol Biol. 2003 Jun;12(3):241-5. doi: 10.1046/j.1365-2583.2003.00407.x. PMID 12752657
- [Background] Hill N, Zhou HN, Wang P, Guo X, Carneiro I, Moore SJ. A household randomized, controlled trial of the efficacy of 0.03% transfluthrin coils alone and in combination with long-lasting insecticidal nets on the incidence of Plasmodium falciparum and Plasmodium vivax malaria in Western Yunnan Province, China. Malar J. 2014 May 31;13:208. doi: 10.1186/1475-2875-13-208. PMID 24885993
- [Background] Kawada H, Temu EA, Minjas JN, Matsumoto O, Iwasaki T, Takagi M. Field evaluation of spatial repellency of metofluthrin-impregnated plastic strips against Anopheles gambiae complex in Bagamoyo, coastal Tanzania. J Am Mosq Control Assoc. 2008 Sep;24(3):404-9. doi: 10.2987/5743.1. PMID 18939693
- [Background] Keita M, Traore S, Sogoba N, Dicko AM, Coulibaly B, Sacko A, Doumbia S, Traore SF. [Susceptibility status of Anopheles gambiae sensu lato to insecticides commonly used for malaria control in Mali]. Bull Soc Pathol Exot. 2016 Feb;109(1):39-45. doi: 10.1007/s13149-015-0461-2. Epub 2016 Jan 6. French. PMID 26740098
- [Background] Lucas JR, Shono Y, Iwasaki T, Ishiwatari T, Spero N, Benzon G. U.S. laboratory and field trials of metofluthrin (SumiOne) emanators for reducing mosquito biting outdoors. J Am Mosq Control Assoc. 2007 Mar;23(1):47-54. doi: 10.2987/8756-971X(2007)23[47:ULAFTO]2.0.CO;2. PMID 17536367
- [Background] Ogoma SB, Moore SJ, Maia MF. A systematic review of mosquito coils and passive emanators: defining recommendations for spatial repellency testing methodologies. Parasit Vectors. 2012 Dec 7;5:287. doi: 10.1186/1756-3305-5-287. PMID 23216844
- [Background] Syafruddin D, Bangs MJ, Sidik D, Elyazar I, Asih PB, Chan K, Nurleila S, Nixon C, Hendarto J, Wahid I, Ishak H, Bogh C, Grieco JP, Achee NL, Baird JK. Impact of a spatial repellent on malaria incidence in two villages in Sumba, Indonesia. Am J Trop Med Hyg. 2014 Dec;91(6):1079-87. doi: 10.4269/ajtmh.13-0735. Epub 2014 Oct 13. PMID 25311699
- [Background] Tripet F, Wright J, Cornel A, Fofana A, McAbee R, Meneses C, Reimer L, Slotman M, Thiemann T, Dolo G, Traore S, Lanzaro G. Longitudinal survey of knockdown resistance to pyrethroid (kdr) in Mali, West Africa, and evidence of its emergence in the Bamako form of Anopheles gambiae s.s. Am J Trop Med Hyg. 2007 Jan;76(1):81-7. PMID 17255234
- [Derived] Van Hulle S, Sagara I, Mbodji M, Nana GI, Coulibaly M, Dicko A, Kone M, Thera I, Sylla D, Traore MD, Liu F, Grieco JP, Achee NL. Evaluation of the protective efficacy of a spatial repellent to reduce malaria incidence in children in Mali compared to placebo: study protocol for a cluster-randomized double-blinded control trial (the AEGIS program). Trials. 2022 Apr 5;23(1):259. doi: 10.1186/s13063-022-06197-w. PMID 35382856
- See also: Demographic Health Survey, Mali, 2018 — https://dhsprogram.com/pubs/pdf/SR261/SR261.E.pdf
- See also: Demographic Health Survey, Mali, 2015 — https://dhsprogram.com/what-we-do/survey/survey-display-487.cfm
- See also: Health Management Information System, DHIS2, 2018 — https://www.dhis2.org/about
- See also: Recensement General de la Population et de l'Habitat du Mali (RGPH) 2009 — https://catalog.ihsn.org/index.php/catalog/4569